CLINICAL TRIAL: NCT03057873
Title: A Double Blind, Placebo Controlled Parallel Study to Investigate the Effect of a High Protein, High Fiber Dietary Supplement on Weight and Fat Loss in Healthy Overweight Adults
Brief Title: The Effect of a High Protein, High Fiber Dietary Supplement on Weight and Fat Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beachbody (Industry)
Collaborators: KGK Science Inc. (Industry); Glycemic Index Laboratories, Inc (Industry); MB Clinical Research and Consulting LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 15SWHB
Record Dates: First submitted 2017-02-16; First posted 2017-02-20 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Overweight
Keywords: protein; fiber; weight loss; fat loss
MeSH Terms: conditions — Overweight; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High protein, high fiber (Experimental): Participants receive a high protein, high fiber dietary supplement twice daily (30 minutes before breakfast and lunch) for 12 weeks
  Interventions: Dietary Supplement: High protein, high fiber dietary supplement
- Low protein, low fiber (Placebo Comparator): Participants receive a low protein, low fiber supplement twice daily (30 minutes before breakfast and lunch) for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: High protein, high fiber dietary supplement — Dry powder to be mixed with 10 ounces of cold water
  Arms: High protein, high fiber
Dietary Supplement: Placebo — Dry powder to be mixed with 10 ounces of cold water
  Arms: Low protein, low fiber

SUMMARY:
The objective of this study is to investigate the effect of a high protein, high fiber dietary supplement on weight and fat loss in healthy overweight adults. Half of participants will receive a high protein, high fiber supplement twice a day for 12 weeks, and half of the subjects will receive a placebo (that contains the same amount of calories as the supplement) twice a day for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of 25-50 years of age
2. If female, the subject is not of child bearing potential, which is defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation) OR

   Females of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result at screening. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System) for at least 3 months
   * Double-barrier method
   * Non-hormonal IUDs
   * Hormonal IUD methods must be a stable dose for at least 3 months
   * Vasectomy of partner
   * Non-heterosexual lifestyle
3. A BMI between 27.0 - <35.0 kg/m2 (inclusive). Subjects must meet exactly the inclusion BMI at screening, or be screen failed. Subjects who meet the BMI requirement at screening and present at run-in with a BMI of <27.0 or >35 kg/m2 will be counselled.
4. Subjects that have had a stable weight for the past 6 months. A stable weight is defined as not having gained or lost more than 5 kg of body weight throughout the past 6 months (cycling of weight, for example, continuously up and down anything less than 5 kg is considered stable)
5. Agreement to comply with dietary recommendations from nutritionist throughout the duration of the study that include a 500 kcal energy deficit from their predicted total energy requirements
6. Agrees to fully comply with all study procedures
7. Has given voluntary written and informed consent to participate in the study
8. Determined to be healthy as per laboratory parameters and physical examination

Exclusion Criteria:

1. Females who are pregnant, breastfeeding or planning to become pregnant during the course of the study
2. Subjects who are smokers (tobacco, e-cigarettes) or have been a smoker within the past 1 year from screening
3. Individuals who carry an epi-pen, or those with a diagnosed allergy or who believe that they have an allergy to milk or milk products, crustacean shellfish, tree nuts, or peanuts
4. Individuals with a severe allergy to egg, fish, wheat or soy ingredients as the product is manufactured in a facility that contains these ingredients
5. The use of prescription, over-the-counter health products, or natural health products/dietary supplements being taken for weight loss, cholesterol levels, or blood pressure within 4 weeks of screening
6. Subjects with a history of eating disorders
7. Current participation or participation within the last 3 months in any weight loss program or diet (for example Weight Watchers, Jenny Craig, DASH diet, Atkins, Mediterranean etc.)
8. Medical history of thyroid disorders except for subjects diagnosed with hypothyroid and have been on stable medication for at least the last 3 months prior to enrollment. All subject with medical history of hyperthyroid are excluded
9. Medical history of hypercholesterolipidemia
10. Use of cholesterol lowering prescription drugs within the last 6 months
11. Fasting TGs ≥ 200 mg/dL (2.26 mmol/L) or a fasting total cholesterol ≥ 240 mg/dL (6.216 mmol/L)
12. Fasting glucose ≥ 126 mg/dL
13. Hypertension defined as untreated systolic blood pressure >160 mmHg, diastolic blood pressure >100 mmHg, or the use of prescription high blood pressure/hypertension medications within the last 6 months
14. Type I or Type II diabetes or use of diabetes medication in a preventative setting.
15. History of gastrointestinal dysfunction or surgery that may influence digestion or absorption
16. Chronic inflammation or structural abnormality, including history of, of the digestive tract (inflammatory bowel disease, celiac disease, chronic diarrhea, chronic constipation, duodenal or gastric ulcer, gastric retention or obstruction, Gastroesophageal reflux disease (GERD), or symptomatic cholelithiasis)
17. Subjects who have a history of colorectal cancer, bowel resection, rectocele, or colostomy
18. Immunocompromised individuals such as subjects that have undergone organ transplantation, those with rheumatoid arthritis, or subjects diagnosed with human immunodeficiency virus (HIV)
19. Unstable medical conditions that in the opinion of the Qualified Investigator preclude the subject from participating in the study
20. Anti-anxiety and anti-psychotic medications will be assessed by the MD on a case by case basis
21. Alcohol use > 2 standard alcoholic drinks per day
22. Alcohol or drug abuse within the last 6 months
23. Use of medicinal marijuana
24. Cancer, except skin cancers completely excised with no chemotherapy or radiation with a follow up that is negative
25. Subjects with metal fixation plates or screws from a previous surgery
26. Clinically significant abnormal laboratory results at screening
27. Participation in a clinical research trial within 30 days prior to randomization
28. Allergy or sensitivity to study supplement ingredients
29. Individuals who are cognitively impaired and/or who are unable to give informed consent
30. Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject
31. Unwilling or unable to comply with study timeline and procedures
32. Individuals who do not like the taste of chocolate or shake type drinks

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 206 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

PRIMARY OUTCOMES:
Change in body weight (kg) | Baseline and 12 weeks
  Body weight measured by clinic study staff at required visits
Change in body fat percentage (%) | Baseline and 12 weeks
  Body fat percentage as determined by dual x-ray absorptiometry (DXA)

SECONDARY OUTCOMES:
Change in total fat mass (kg) | Baseline and 12 weeks
  Body fat mass as determined by DXA
Change in total lean mass (kg) | Baseline and 12 weeks
  Body lean mass as determined by DXA
Change in percent abdominal fat (%) | Baseline and 12 weeks
  Abdominal fat percentage as determined by DXA
Change in percent android fat (%) | Baseline and 12 weeks
  Android fat percentage as determined by DXA
Change in percent gynoid fat (%) | Baseline and 12 weeks
  Gynoid fat percentage as determined by DXA
Change in percent trunk fat (%) | Baseline and 12 weeks
  Trunk fat percentage as determined by DXA
Change in percent leg fat (%) | Baseline and 12 weeks
  Leg fat percentage as determined by DXA
Change in body weight (kg) | Baseline and 4 weeks
  Body weight measured by clinic study staff at required visits
Change in body weight (kg) | Baseline and 8 weeks
  Body weight measured by clinic study staff at required visits
Change in Waist circumference (cm) | Baseline and 4 weeks
  measured with a tape measure at the part of the trunk located midway between the lower costal margin and the iliac crest while the person is standing
Change in Waist circumference (cm) | Baseline and 8 weeks
  measured with a tape measure at the part of the trunk located midway between the lower costal margin and the iliac crest while the person is standing
Change in Waist circumference (cm) | Baseline and 12 weeks
  measured with a tape measure at the part of the trunk located midway between the lower costal margin and the iliac crest while the person is standing
Change in Hip circumference (cm) | Baseline and 4 weeks
  measured with a tape measure around the greater trochanteric prominence (the widest part of the hips)
Change in Hip circumference (cm) | Baseline and 8 weeks
  measured with a tape measure around the greater trochanteric prominence (the widest part of the hips)
Change in Hip circumference (cm) | Baseline and 12 weeks
  measured with a tape measure around the greater trochanteric prominence (the widest part of the hips)
Change in Waist to hip ratio | Baseline and 4 weeks
  Ratio of waist circumference to hip circumference
Change in Waist to hip ratio | Baseline and 8 weeks
  Ratio of waist circumference to hip circumference
Change in Waist to hip ratio | Baseline and 12 weeks
  Ratio of waist circumference to hip circumference
Change in Blood leptin (ng/mL) | Baseline and 12 weeks
  Fasting level of leptin in the blood
Change in Blood adiponectin (mcg/mL) | Baseline and 12 weeks
  Fasting level of adiponectin in the blood
Change in Total cholesterol (mg/dL) | Baseline and 4 weeks
  Fasting level of total cholesterol in blood
Change in Total cholesterol (mg/dL) | Baseline and 8 weeks
  Fasting level of total cholesterol in blood
Change in Total cholesterol (mg/dL) | Baseline and 12 weeks
  Fasting level of total cholesterol in blood
Change in low-density lipoprotein (LDL) Cholesterol (mg/dL) | Baseline and 4 weeks
  Fasting level of LDL cholesterol in blood
Change in low-density lipoprotein (LDL) Cholesterol (mg/dL) | Baseline and 8 weeks
  Fasting level of LDL cholesterol in blood
Change in low-density lipoprotein (LDL) Cholesterol (mg/dL) | Baseline and 12 weeks
  Fasting level of LDL cholesterol in blood
Change in high-density lipoprotein (HDL) Cholesterol (mg/dL) | Baseline and 4 weeks
  Fasting level of HDL cholesterol in blood
Change in high-density lipoprotein (HDL) Cholesterol (mg/dL) | Baseline and 8 weeks
  Fasting level of HDL cholesterol in blood
Change in high-density lipoprotein (HDL) Cholesterol (mg/dL) | Baseline and 12 weeks
  Fasting level of HDL cholesterol in blood
Change in oxidized LDL (Ox-LDL) Cholesterol (U/L) | Baseline and 4 weeks
  Fasting level of Ox-LDL cholesterol in blood
Change in oxidized LDL (Ox-LDL) Cholesterol (U/L) | Baseline and 8 weeks
  Fasting level of Ox-LDL cholesterol in blood
Change in oxidized LDL (Ox-LDL) Cholesterol (U/L) | Baseline and 12 weeks
  Fasting level of Ox-LDL cholesterol in blood
Change in triglycerides (mg/dL) | Baseline and 4 weeks
  Fasting level of triglycerides in blood
Change in triglycerides (mg/dL) | Baseline and 8 weeks
  Fasting level of triglycerides in blood
Change in triglycerides (mg/dL) | Baseline and 12 weeks
  Fasting level of triglycerides in blood
Change in Insulin (IU) | Baseline and 4 weeks
  Fasting level of insulin in blood
Change in Insulin (IU) | Baseline and 8 weeks
  Fasting level of insulin in blood
Change in Insulin (IU) | Baseline and 12 weeks
  Fasting level of insulin in blood
Change in Glucose (mmol/L) | Baseline and 4 weeks
  Fasting level of glucose in blood
Change in Glucose (mmol/L) | Baseline and 8 weeks
  Fasting level of glucose in blood
Change in Glucose (mmol/L) | Baseline and 12 weeks
  Fasting level of glucose in blood
Change in blood glycated haemoglobin (HbA1c) (mmol/mol) | Baseline and 12 weeks
  Fasting level of HbA1c in blood
Change in gut microbiota composition | Baseline and 12 weeks
  Genera of bacteria measured in stool samples

OTHER OUTCOMES:
Change in Modified Gastrointestinal Symptoms Rating Scale (GSRS) dimensions | Baseline and 4 weeks
  Score on each of the 6 dimensions contained in the validated Modified GSRS tool (scores 1-7)
Change in Modified Gastrointestinal Symptoms Rating Scale (GSRS) dimensions | Baseline and 8 weeks
  Score on each of the 6 dimensions contained in the validated Modified GSRS tool (scores 1-7)
Change in Modified Gastrointestinal Symptoms Rating Scale (GSRS) dimensions | Baseline and 12 weeks
  Score on each of the 6 dimensions contained in the validated Modified GSRS tool (scores 1-7)
Change in Bowel Habits (number of bowel movements/day; Bristol Stool form type) | Baseline and 4 weeks
  Bowel habits assessed for 72-hour period every 2 weeks by bowel habits diary including number of bowel movements per day and classification of stool form type. Data for each time point (4, 8, and 12 weeks) will include 2 diary collections.
Change in Bowel Habits (number of bowel movements/day; Bristol Stool form type) | Baseline and 8 weeks
  Bowel habits assessed for 72-hour period every 2 weeks by bowel habits diary including number of bowel movements per day and classification of stool form type. Data for each time point (4, 8, and 12 weeks) will include 2 diary collections.
Change in Bowel Habits (number of bowel movements/day; Bristol Stool form type) | Baseline and 12 weeks
  Bowel habits assessed for 72-hour period every 2 weeks by bowel habits diary including number of bowel movements per day and classification of stool form type. Data for each time point (4, 8, and 12 weeks) will include 2 diary collections.
Change in systolic blood pressure | Baseline and 4 weeks
  Seated resting blood pressure will be determined from 3 measurements obtained at least 1 minute apart
Change in systolic blood pressure | Baseline and 8 weeks
  Seated resting blood pressure will be determined from 3 measurements obtained at least 1 minute apart
Change in systolic blood pressure | Baseline and 12 weeks
  Seated resting blood pressure will be determined from 3 measurements obtained at least 1 minute apart
Change in diastolic blood pressure | Baseline and 4 weeks
  Seated resting blood pressure will be determined from 3 measurements obtained at least 1 minute apart
Change in diastolic blood pressure | Baseline and 8 weeks
  Seated resting blood pressure will be determined from 3 measurements obtained at least 1 minute apart
Change in diastolic blood pressure | Baseline and 12 weeks
  Seated resting blood pressure will be determined from 3 measurements obtained at least 1 minute apart
Change in Profiles of Mood States (POMS) questionnaire ratings | Baseline and 4 weeks
  Scores for energy, mood, and stress as assessed by POMS questionnaire
Change in Profiles of Mood States (POMS) questionnaire ratings | Baseline and 8 weeks
  Scores for energy, mood, and stress as assessed by POMS questionnaire
Change in Profiles of Mood States (POMS) questionnaire ratings | Baseline and 12 weeks
  Scores for energy, mood, and stress as assessed by POMS questionnaire
Change in Three-factor Eating Questionnaire (TFEQ) scores | Baseline and 4 weeks
  Scores for eating behavior as assessed by TFEQ
Change in Three-factor Eating Questionnaire (TFEQ) scores | Baseline and 8 weeks
  Scores for eating behavior as assessed by TFEQ
Change in Three-factor Eating Questionnaire (TFEQ) scores | Baseline and 12 weeks
  Scores for eating behavior as assessed by TFEQ
Change in Binge Eating Scale (BES) scores | Baseline and 4 weeks
  Scores for binge eating as assessed by BES
Change in Binge Eating Scale (BES) scores | Baseline and 8 weeks
  Scores for binge eating as assessed by BES
Change in Binge Eating Scale (BES) scores | Baseline and 12 weeks
  Scores for binge eating as assessed by BES
Change in number of junk food cravings reported | Baseline and 4 weeks
  Number of cravings as assessed by daily entries in study diary
Change in number of junk food cravings reported | Baseline and 8 weeks
  Number of cravings as assessed by daily entries in study diary
Change in number of junk food cravings reported | Baseline and 12 weeks
  Number of cravings as assessed by daily entries in study diary
Change in IgG levels | Baseline and 12 weeks
  Fasting level of IgG in blood
Change in IgA levels | Baseline and 12 weeks
  Fasting level of IgA in blood
Change in IgM levels | Baseline and 12 weeks
  Fasting level of IgM in blood
Change in Complement C3 levels | Baseline and 12 weeks
  Fasting level of C3 in blood
Change in Complement C4 levels | Baseline and 12 weeks
  Fasting level of C4 in blood

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.; Thomas Wolever, MD, PhD, Principal Investigator — Glycemic Index Laboratories, Inc; Rupal Trivedi, MD, Principal Investigator — Great Lakes Clinical Trials (of MB Clinical Research and Consulting, LLC)
Locations (3):
- Great Lakes Clinical Trials (of MB Clinical Research and Consulting, LLC), Chicago, Illinois, United States
- Canada (2):
  - KGK Synergize Inc., London, Ontario
  - GI Labs, Inc., Toronto, Ontario

REFERENCES:
- [Derived] Glynn EL, Fleming SA, Edwards CG, Wilson MJ, Evans M, Leidy HJ. Consuming a Protein and Fiber-Based Supplement Preload Promotes Weight Loss and Alters Metabolic Markers in Overweight Adults in a 12-Week, Randomized, Double-Blind, Placebo-Controlled Trial. J Nutr. 2022 Jun 9;152(6):1415-1425. doi: 10.1093/jn/nxac038. PMID 35212740